CLINICAL TRIAL: NCT05812365
Title: Best End-Expiratory and Driving-Pressure for Individualized Flow Controlled Ventilation in Patients With COPD - an Observational Study.
Brief Title: Best End-Expiratory and Driving-pressure for Individualized Flow Controlled Ventilation in Patients With COPD
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Ventinova Medical, Eindhoven, Netherlands (Unknown); Timple SA, Rua Simao Álvares 356 Conj. 41,42 e 51 - Pinheiros, Sao Paulo (Brasilien) (Unknown)
Responsible Party: Principal Investigator, André Dankert, MD, Principal Investigator, Universitätsklinikum Hamburg-Eppendorf
Other Study IDs: 2023-101013
Record Dates: First submitted 2023-04-02; First posted 2023-04-13 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: COPD; Ventilator Lung; Anesthesia
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with chronic obstructive pulmonary disease (COPD) have a significantly increased risk of postoperative pulmonary complications (PPC). Protective ventilation of the lungs could reduce the rate of PPC in patients with COPD. It has been suggested that flow controlled ventilation (FCV) may be less invasive and more protective to the lungs than conventional ventilation in patients with COPD.

The primary aim of this study is to determine a optimal individual ventilation setting for FCV in ten participants with COPD.

DETAILED DESCRIPTION:
The estimated worldwide chronic obstructive pulmonary disease (COPD) mean prevalence is 13.1%. In 2015, 3.2 million people died from COPD worldwide, and estimates show that COPD will be the third leading cause of death in 2030. Patients with COPD are at high risk for postoperative pulmonary complications (PPC). It has been proposed that FCV might be less-invasive and more protective for the lungs than conventional ventilation in patients with COPD. The pathophysiology of COPD is multifactorial, with the collapse of the central airways having a major impact on the symptoms. Minimizing the expiratory flow could prevent this airway pathology, and thus be beneficial in the ventilation of patients with COPD.

In the operation theater participants will be ventilated with flow controlled ventilation (FCV). Arterial blood gas analysis and electrical impedance tomography (EIT) will be measured.

The aim of the study is to determine the best end-expiratory pressure and driving pressure (assessed after anesthesia induction based on compliance and EIT parameters).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing surgery with endotracheal intubation
* Age ≥ 18
* Verified COPD (preoperative spirometry)

Exclusion Criteria:

* Pregnant woman
* Laparoscopic surgery
* Surgery that might interfere with EIT measurement
* Cardiac Implantable Electronic Devices

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with verified COPD, scheduled for operations in general anesthesia, who present in the preassessment clinic of the University Medical Center Hamburg-Eppendorf during the study recruitment period, will be screened for eligibility.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-07-24 (Actual); Study Completion 2024-07-24 (Actual)

PRIMARY OUTCOMES:
Best end-expiratory pressure | 1 hour after tracheal Intubation
  Best end-expiratory pressure (mbar), defined as the end-expiratory pressure associated with the best compliance, best tradeoff between alveolar collapse and hyper distension (EIT)

SECONDARY OUTCOMES:
Best driving pressure | 1 hour after tracheal intubation
  Best driving pressure (peek pressure - end-expiratory pressure in mbar) associated with the best compliance, best tradeoff between alveolar collapse and hyper distension (EIT)
Dissipated energy | 1 hour after tracheal intubation
  Calculated dissipated energy per liter of gas ventilated (J) during ventilation.
Required minute volume to maintain carbon dioxide partial pressure (pCO2) level | 1 hour after tracheal intubation
  The minute volume (L/min) of the ventilator will be adjusted to maintain the preoperative baseline pCO2 level (blood gas analysis).
Applied mechanical power | 1 hour after tracheal intubation
  Calculated applied mechanical power during ventilation (J/min)
Ventilation distribution | 1 hour after tracheal intubation
  Expressed as the percentage of total pulmonary ventilation through each of the regions-of-interest, total 100%.
Delta Z | 1 hour after tracheal intubation
  Measured variation of impedance (arbitrary units) by electrical impedance tomography.
Delta end-expiratory lung impedance | 1 hour after tracheal intubation
  Variation of impedance plethysmography at end-expiration measured by electrical impedance tomography.
Distribution of regional tidal ventilation | 1 hour after tracheal intubation
  Distribution of regional tidal ventilation will be determined as the relation of regional ΔZ/total ΔZ (expressed in percentage), measured by electrical impedance tomography.
Regional lung compliance | 1 hour after tracheal intubation
  Calculated by electrical impedance tomography (ml/cm H2O)
Center of Ventilation | 1 hour after tracheal intubation
  Variations of the pulmonary ventilation distribution in the ventral-dorsal and left-right direction measured by electrical impedance tomography.
Global inhomogeneity index | 1 hour after tracheal intubation
  Impedance variations of each pixel between the end of inspiration and expiration measured by electrical impedance tomography.
arterial oxygen partial pressure (paO2) | 1 hour after tracheal intubation
  Measured by blood gas analysis (mmHg)
carbon dioxide partial pressure (pCO2) | 1 hour after tracheal intubation
  Measured by blood gas analysis (mmHg)
Horovitz quotient | 1 hour after tracheal intubation
  Ratio of PaO2 (mmHg) and the fraction of oxygen of the inhaled air (FiO2).
Base excess | 1 hour after tracheal intubation
  Measured by blood gas analysis (mmol/l)
potential of hydrogen (pH) | 1 hour after tracheal intubation
  Measured by blood gas analysis
Resistance | 1 hour after tracheal intubation
  Pressure change per flow change measured by the ventilator (kPa*s/l).
tidal volume | 1 hour after tracheal intubation
  Measure by ventilator (ml)
Peak inspiratory pressure | 1 hour after tracheal intubation
  Maximum pressure during the inspiration measured by the ventilator (mbar).
Respiratory rate | 1 hour after tracheal intubation
  Measured by the ventilator (1/min)
End-tidal carbon dioxide (etCO2) | 1 hour after tracheal intubation
  End-tidal carbon dioxide level measured by the ventilator (mmHg).

CONTACTS AND LOCATIONS:
Overall Officials: André Dankert, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf; Martin Petzoldt, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blanco I, Diego I, Bueno P, Casas-Maldonado F, Miravitlles M. Geographic distribution of COPD prevalence in the world displayed by Geographic Information System maps. Eur Respir J. 2019 Jul 18;54(1):1900610. doi: 10.1183/13993003.00610-2019. Print 2019 Jul. No abstract available. PMID 31000678
- [Background] GBD 2015 Chronic Respiratory Disease Collaborators. Global, regional, and national deaths, prevalence, disability-adjusted life years, and years lived with disability for chronic obstructive pulmonary disease and asthma, 1990-2015: a systematic analysis for the Global Burden of Disease Study 2015. Lancet Respir Med. 2017 Sep;5(9):691-706. doi: 10.1016/S2213-2600(17)30293-X. Epub 2017 Aug 16. PMID 28822787
- [Background] Mathers CD, Loncar D. Projections of global mortality and burden of disease from 2002 to 2030. PLoS Med. 2006 Nov;3(11):e442. doi: 10.1371/journal.pmed.0030442. PMID 17132052
- [Background] Dankert A, Neumann-Schirmbeck B, Dohrmann T, Greiwe G, Plumer L, Loser B, Sehner S, Zollner C, Petzoldt M. Preoperative Spirometry in Patients With Known or Suspected Chronic Obstructive Pulmonary Disease Undergoing Major Surgery: The Prospective Observational PREDICT Study. Anesth Analg. 2023 Oct 1;137(4):806-818. doi: 10.1213/ANE.0000000000006235. Epub 2022 Nov 1. PMID 36730893
- [Background] Tsuboi N, Tsuboi K, Nosaka N, Nishimura N, Nakagawa S. The Ventilatory Strategy to Minimize Expiratory Flow Rate in Ventilated Patients with Chronic Obstructive Pulmonary Disease. Int J Chron Obstruct Pulmon Dis. 2021 Feb 12;16:301-304. doi: 10.2147/COPD.S296343. eCollection 2021. PMID 33603356
- [Background] Barnes T, van Asseldonk D, Enk D. Minimisation of dissipated energy in the airways during mechanical ventilation by using constant inspiratory and expiratory flows - Flow-controlled ventilation (FCV). Med Hypotheses. 2018 Dec;121:167-176. doi: 10.1016/j.mehy.2018.09.038. Epub 2018 Sep 24. PMID 30396474
- [Background] Bauer M, Opitz A, Filser J, Jansen H, Meffert RH, Germer CT, Roewer N, Muellenbach RM, Kredel M. Perioperative redistribution of regional ventilation and pulmonary function: a prospective observational study in two cohorts of patients at risk for postoperative pulmonary complications. BMC Anesthesiol. 2019 Jul 27;19(1):132. doi: 10.1186/s12871-019-0805-8. PMID 31351452
- [Background] Borges JB, Cronin JN, Crockett DC, Hedenstierna G, Larsson A, Formenti F. Real-time effects of PEEP and tidal volume on regional ventilation and perfusion in experimental lung injury. Intensive Care Med Exp. 2020 Feb 21;8(1):10. doi: 10.1186/s40635-020-0298-2. PMID 32086632
- [Background] Dankert A, Dohrmann T, Loser B, Zapf A, Zollner C, Petzoldt M. Pulmonary Function Tests for the Prediction of Postoperative Pulmonary Complications. Dtsch Arztebl Int. 2022 Feb 18;119(7):99-106. doi: 10.3238/arztebl.m2022.0074. PMID 34939921